CLINICAL TRIAL: NCT03076892
Title: A Phase II Study Evaluating the Non-inferiority and Better Tolerability of the Device PHOS-ISTOS Compared to the Conventional Photodynamic Therapy (PDT)
Brief Title: Evaluation of Non-inferiority and Tolerability of the Device PHOS-ISTOS
Acronym: PHOS-ISTOS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Collaborators: European Commission (Other); Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2015_79; 2016-A00010-51 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2017-03-07; First posted 2017-03-10 (Actual); Last update posted 2017-11-14 (Actual); Status verified 2017-11

CONDITIONS: Keratosis, Actinic
Keywords: PDT; Methyl Aminolevulinate; light emitting textile
MeSH Terms: conditions — Keratosis, Actinic

STUDY DESIGN:
Intervention Model Description: Split Face intra individual comparison
Oversight: Data Monitoring Committee: No

ARMS (2):
- Conventional PDT (Active Comparator): Aktilite® Galderma
  Interventions: Device: Aktilite® Galderma
- PHOS ISTOS PDT (Experimental): Light Emitting textile device
  Interventions: Device: PHOS ISTOS PDT

INTERVENTIONS:
Device: Aktilite® Galderma — preparation of the lesions, Metvixia application + occlusive dressing during 3 hours + illumination: 7 to 10 minutes
  Other Names: Conventional PDT
  Arms: Conventional PDT
Device: PHOS ISTOS PDT — preparation of the lesions, Metvixia application + occlusive dressing during 30 minutes + illumination: 2.5 hours
  Arms: PHOS ISTOS PDT

SUMMARY:
This study aims to compare the efficacy and tolerance of a new photodynamic therapy device (PHOS-ISTOS) with the conventional PDT device (Aktilite®) for the treatment of actinic keratosis of the scalp

DETAILED DESCRIPTION:
The study is an intraindividual comparison of two methods. The number of subjects to be enrolled is 47. Patients will receive both treatments in a single visit: A first period of 2.5 hours of illumination with Phos-Istos device followed by a continuous red light spectrum (between 7 and 10 minutes) with Aktilite® after an appropriate incubation of MAL (methyl aminolevulinate). Patients will complete a pain assessment scale after receiving both treatments. 3 follow-up visits will be then scheduled

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of minimum 10 previously untreated not pigmented, non-hyperkeratotic AK lesions of Grade I and II of the forehead and/or scalp (according to Olsen et Al. JAAD 1991, cf. REF 31) where other therapies are unacceptable or considered medically less appropriate with a symmetrical repartition on both side of the forehead and/or scalp. The diagnosis of AK will be determined upon clinical evaluation (i.e. visual inspection and palpation) by the investigator.
* No treatment for the AKs in the previous 30 days.
* Symmetrical areas in terms of number and severity of lesions. The axis of symmetry between the two areas will be defined by the investigator according to the distribution of lesions.
* The two areas to be treated should not be coalescing. A minimum distance of 10 mm is required between the lesions located on the 2 symmetrical areas. A minimum distance of 2 mm is required between the lesions on the same side.
* Minimum 5 lesions with similar dimensions at both symmetrical areas will be treated. If the number of lesions is >7, only 7 lesions on each side will be considered.

Exclusion Criteria:

* Patients with porphyria.
* Patients immunosuppressed for idiopathic, disease specific or therapeutic reasons.
* Use of topical corticosteroids to lesional areas within 2 weeks before PDT.
* Patients receiving local treatment (including cryotherapy and curettage-electrocoagulation, any PDT treatment) in face / scalp area within the last 30 days.
* Patients receiving topical treatment (including imiquimod, 5-FU and diclofenac, Picato) in face / scalp area within the last 30 days.in
* Use of topical retinoids or alpha-hydroxy acids, systemic retinoids, chemotherapy or immunotherapy within 30 days of PDT.
* Pigmented AK lesion(s).
* Known allergy to Metvixia/Metvix, a similar PDT compound or excipients of the cream including arachis oil, or to peanut or soya.
* Participation in other clinical studies either currently or within the last 30 days.
* Female subjects must be of either:

  * Non-childbearing potential, i.e. post-menopausal or have a confirmed clinical history of sterility (e.g. the subject is without a uterus) or,
  * Childbearing potential, provided there is a confirmed negative urine pregnancy test or blood analysis prior to study treatment, to rule out pregnancy.
* Any condition which may be associated with a risk of poor protocol compliance.
* Patients currently receiving regular ultraviolet radiation therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2017-11 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Treated lesion response rate | up to Month 6
  Each treatment area will be counted, graded with Clinical grade of AK, mapped and photographed

SECONDARY OUTCOMES:
Visual analog scale of pain | at Day 1 and Day 7
  measure the pain and local tolerance graduation range 0 to 10.
Scale for clinical assessment of the subject's skin aspect | at Month 3 and Month 6
  4-point scale that ranged of Excellent :No scarring, atrophy or induration, and no or slight occurrence of redness or change in pigmentation compared to adjacent skin Good: No scarring, atrophy or induration but moderate redness or change in pigmentation compared to adjacent skin Fair: Slight to moderate occurrence of scarring, atrophy or induration Poor : Extensive occurrence of scarring, atrophy or induration
Rate of patients with at least 75% of reduction of the lesions | at Month 3 and Month 6
  The response rate is calculated in relation to the initial number of lesions: Response rate is validated if rate ≥ 4 lesions destroyed for 5 initial lesions, ≥ 5 for 6 lesions and ≥ 6 for 7 lesions
Dermatology Life Quality Index (DLQI ) | at day 1 , Day 7, Month 3 and Month 6
  The questionnaire of 10 questions is completed by the patient to evaluate his quality of life
Satisfaction autoquestionnaire | at Day 7, Month 3 and Month 6
  The questionnaire is created by investigator to evaluate the comfort of device.
  Participants will answer 9 questions on a 5-point scale that ranged from Not embarrassing,few embarrassing, Embarrassing, Very embarrassing, Don't know

CONTACTS AND LOCATIONS:
Overall Officials: Laurent Mortier, MD, PhD, Principal Investigator — University Hospital, Lille
Locations (2):
- CHRU, Hôpital Claude Huriez, Lille, France
- Klinikum Vest Gmbh, Recklinghausen, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Vignion-Dewalle AS, Abi Rached H, Thecua E, Lecomte F, Deleporte P, Behal H, Hommel T, Duhamel A, Szeimies RM, Mortier L, Mordon S. A New Light-Emitting, Fabric-Based Device for Photodynamic Therapy of Actinic Keratosis: Protocol for a Randomized, Controlled, Multicenter, Intra-Individual, Phase II Noninferiority Study (the Phosistos Study). JMIR Res Protoc. 2019 Apr 26;8(4):e12990. doi: 10.2196/12990. PMID 31025953